CLINICAL TRIAL: NCT06491862
Title: RACE-2L: Real-World Assessment of Clinical Practice and Outcomes in Non-squamous Non-Small Cell Lung Cancer After Failure of Platinum-based Chemotherapy in Brazil
Brief Title: RACE-2L: Real-World Assessment of Clinical Practice and Outcomes in Non-squamous NSCLC After Failure of Platinum-based Chemotherapy in Brazil
Acronym: RACE-2L
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133HR00041
Record Dates: First submitted 2024-06-11; First posted 2024-07-09 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Non-squamous Non-Small Cell Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will be implemented as a retrospective, noninterventional medical record review of patients from routine practice settings who have been diagnosed with a/m non-squamous NSCLC with or without AGA and received at least 1 line of systemic treatment after failing PTC between January 2017 and December 2024.

DETAILED DESCRIPTION:
The study will be implemented as a retrospective, noninterventional medical record review of patients from routine practice settings who have been diagnosed with advanced/metastaic non-squamous NSCLC with or without AGA and who have failed platinum-based chemotherapy and immunotherapy (for patients without AGA) or platinum-based chemotherapy and at least 1 line of targeted therapy (for patients with AGA). The study will be conducted on one cohort of patients regardless their AGA status. The study index date will be defined as first dose of any agent after PTC, with specific treatments received for AGA and non-AGA patients in the preindex period. We will also conduct a subgroup analysis on NSCLC pre-defined subtypes (sample size permitting): EGFR mutant, ALK translocation, ROS1 translocation, MET1 mutant, HER-2 mutant, BRAF mutant, pan-wild-type PD-L1 >50%.

ELIGIBILITY:
Inclusion Criteria

* Confirmed diagnosis of patients with non-squamous NSCLC stage IIIB/IIIC not eligible for curative-intent therapies or stage IV/M1 (a/m NSCLC) with or without actionable genomic mutations (i.e., EGFR, ALK, ROS1, NTRK, BRAF, MET exon 14 skipping, RET, HER-2)
* Aged at least 18 years at first diagnosis of a/m NSCLC
* For the AGA subgroup, having received platinum-based chemotherapy, having received at least one target approved therapy.
* For the non_AGA subgroup,should have received either sequential or concurrent use of ICI and PTC)
* Patient must have received at least line of therapy of an active agent after failing PTC.

Exclusion Criteria

* Patients with evidence of other primary malignancies (apart from basal cell carcinoma and melanoma) within 1 year prior to the index date will be excluded from both the study cohorts.
* Patients who participated in an investigational clinical trial for the treatment of any cancer, including NSCLC, or any early access program from 2018 onward.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of sequential adult patients in study sites with a diagnosis of IIIB/IIIC/IV non-squamous NSCLC with or without AGA and received at least 1 line of treatment after failing PTC for a/m NSCLC with a start date between January 2017 and December 2024.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Describe the patient population and treatment patterns | between January 1st 2017 and December 31th 2024
  Description of patient population and treatment patterns: tumor histology, mutation and PD-L1 status, disease stage at diagnosis
Describe the patient population and treatment patterns | between January 1st 2017 and December 21th 2024
  Description of patient population and treatment patterns: disease stage at diagnosis
Describe the patient population and treatment patterns | between January 1st 2017 and December 21th 2024
  Description of patient population and treatment patterns: smoking status
Describe the patient population and treatment patterns | between January 1st 2017 and December 31th 2024
  Description of patient population and treatment patterns: age
Describe the patient population and treatment patterns | between January 1st 2017 and December 31th 2024
  Description of patient population and treatment patterns: gender
Describe the patient population and treatment patterns | between January 1st 2017 and December 31th 2024
  Description of patient population and treatment patterns: presence of brain metastasis at diagnosis
Describe the patient population and treatment patterns | between January 1st 2017 and December 31th 2024
  Description of patient population and treatment patterns: comorbidities (based on Charlson Comorbity Index)
Describe the patient population and treatment patterns | between January 1st 2017 and December 31th 2024
  Description of patient population and treatment patterns: treatments used prior to the index date, their start and end time and response
Describe the patient population and treatment patterns | between January 1st 2017 and December 31th 2024
  Description of patient population and treatment patterns: treatments used after the index date
Describe the patient population and treatment patterns | between January 1st 2017 and December 31th 2024
  Description of patient population and treatment patterns: weight
Describe the patient population and treatment patterns | between January 1st 2017 and December 31th 2024
  Description of patient population and treatment patterns: height
Describe the patient population and treatment patterns | between January 1st 2017 and December 31th 2024
  Description of patient population and treatment patterns: weight change between first treatment for metastatic disease and treatment index
Describe the patient population and treatment patterns | between January 1st 2017 and December 31th 2024
  Description of patient population and treatment patterns: starting dose of the index treatment
Describe of the population and treatment patterns | between January 1st 2017 and December 31th 2024
  Description of patient population and treatment patterns: duration of therapy
Describe the patient population and treatment patterns | between January 1st 2017 and December 31th 2024
  Description of patient population and treatment patterns: reasons for discontinuation

CONTACTS AND LOCATIONS:
Locations (5):
- Brazil (5):
  - Research Site, Belo Horizonte, Minas Gerais
  - Research Site, Natal, Rio Grande do Norte
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, São José do Rio Preto, São Paulo
  - Research Site, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home